CLINICAL TRIAL: NCT02384902
Title: Effect of Dietary Glycemic Index/Load on Kidney-related Biomarkers and Inflammation in Diabetic Nephropathy Patients
Brief Title: Effect of Low GI/ Glycemic Load (GL) Diet in Diabetic Nephropathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Leila Azadbakht, Isfahan University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: low GI nephropathy
Record Dates: First submitted 2014-09-06; First posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Diabetic Nephropathy; Medication Compliance
Keywords: glycemic index; diabetic nephropathy; low glycemic load; inflammation
MeSH Terms: conditions — Diabetic Nephropathies; Medication Adherence; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- low GI (Experimental): low GI: participants were asked to consume low GI foods (GI<55) in abundant, medium GI in moderate and high GI (GI>70) rarely.
  Interventions: Other: low GI
- low GL (Experimental): low GL: participants were asked to consume low GI foods and the amount of carbohydrate was controlled.
  Interventions: Other: low GI
- conventional diet (Experimental): conventional diet: all carbohydrate were treated as the same.
  Interventions: Other: conventional diet

INTERVENTIONS:
Other: low GI — All diets were designed with similar macronutrients content (30% fat, 0.8 g/kg/d protein and remained calorie requirement by carbohydrate). Additionally, we controlled phosphorus, sodium and potassium content of diets for three intervention groups. All dietary menus had less than 1500 mg phosphor and less than 2400 mg sodium and 2000 mg potassium.
  Arms: low GI
Other: low GI — All diets were designed with similar macronutrients content (30% fat, 0.8 g/kg/d protein and remained calorie requirement by carbohydrate). Additionally, we controlled phosphorus, sodium and potassium content of diets for three intervention groups. All dietary menus had less than 1500 mg phosphor and less than 2400 mg sodium and 2000 mg potassium.
  Arms: low GL
Other: conventional diet — All diets were designed with similar macronutrients content (30% fat, 0.8 g/kg/d protein and remained calorie requirement by carbohydrate). Additionally, we controlled phosphorus, sodium and potassium content of diets for three intervention groups. All dietary menus had less than 1500 mg phosphor and less than 2400 mg sodium and 2000 mg potassium.
  Arms: conventional diet

SUMMARY:
low GI and low GL diet have more beneficial effect for diabetic nephropath patients compared with conventional diet.

low GL may have more favorable effect than low GI diet.

DETAILED DESCRIPTION:
According to body weight status of participants, the investigators considered a slight calorie restriction ranged from 200 to 300 Kcal/d. Planed meals and exchange list prescribed for all volunteers. Dietary records forms were given to all subjects and they were educated how to record their dietary intakes. The investigators asked subjects not to change their physical activity level during the study and monitored them for their physical activity level by 3 days physical activity records monthly.

ELIGIBILITY:
Inclusion Criteria:

* diabetic nephropathy, medication stable

Exclusion Criteria:

* poor adherence of dietary recommendations, any changes in kind or dosage of medications

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Serum creatinine (and blood urea nitrogen (BUN) (mg/dL) were measured by colorimetric method and enzymatic colorimetric method using commercial assay kit. | baseline, wk 12

SECONDARY OUTCOMES:
Serum levels of high sensitive C- reactive protein (hs-CRP) (mg/L) were quantified by using an ultrasensitive latex-enhanced immunoturbidimetric assay (Randox Laboratory Ltd., Belfast, United Kingdom). | baseline, wk 12

OTHER OUTCOMES:
Fasting blood sugar (FBS) and lipid profile concentrations (mg/dl) were measured using commercially available enzymatic reagents adopted to an auto-analyzer system. | baseline, wk 12

CONTACTS AND LOCATIONS:
Overall Officials: leila azadbakht, phd, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Leila Azadbakht, Isfahan, Isfahan, Iran